CLINICAL TRIAL: NCT04149262
Title: An Open Label, Single-center, Randomized, Cross-over Trial Comparing the Efficacy and Safety of Faster-acting Insulin Aspart (Fiasp®) Compared to Insulin Aspart (NovoRapid)® Used in the Medtronic MiniMed 640G Insulin Pump Equipped With Sensor
Brief Title: Fiasp® Versus NovoRapid® in Children With Type 1 Diabetes on MiniMed 640G Pump With Sensor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Athanasios Christoforidis, Assistant Professor in Pediatric Endocrinology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AUTH-AC-1
Record Dates: First submitted 2019-10-26; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fiasp/Novorapid (Active Comparator): 4 weeks on Fiasp® then crossover to 4 weeks on NovoRapid® in subjects on the MiniMed 640G system equipped with SmartGuardTM technology and accompanied with EnliteTM Sensor and GuardianTM 2 Link transmitter
  Interventions: Drug: Fiasp; Drug: Novorapid; Device: 640G pump
- Novorapid/Fiasp (Active Comparator): 4 weeks on NovoRapid® then crossover to 4 weeks on Fiasp® in subjects on the MiniMed 640G system equipped with SmartGuardTM technology and accompanied with EnliteTM Sensor and GuardianTM 2 Link transmitter
  Interventions: Drug: Fiasp; Drug: Novorapid; Device: 640G pump

INTERVENTIONS:
Drug: Fiasp — Fiasp® used in a MiniMed 640G system equipped with SmartGuardTM technology and accompanied with EnliteTM Sensor and GuardianTM 2 Link transmitter
Drug: Novorapid — Novorapid® used in a MiniMed 640G system equipped with SmartGuardTM technology and accompanied with EnliteTM Sensor and GuardianTM 2 Link transmitter
Device: 640G pump — MiniMed 640G system equipped with SmartGuardTM technology and accompanied with EnliteTM Sensor and GuardianTM 2 Link

SUMMARY:
This is an exploratory, single-center, open label, randomized, complete cross-over trial comparing safety and efficacy of Fiasp® versus NovoRapid® when used in the Medtronic MiniMed 640G system in pediatric subjects with Type 1 Diabetes Mellitus

DETAILED DESCRIPTION:
This study is designed to compare Fiasp® to NovoRapid® in children with T1DM wearing MiniMed 640G system equipped with SmartGuardTM technology and accompanied with EnliteTM Sensor and GuardianTM 2 Link transmitter in terms of glycemic control with a focus on post-prandial ½-hour and 1-hour plasma glucose levels. The investigator's hypothesis is that post prandial glucoses will be lower and time in range will be greater during the Fiasp® treatment period.

Half, randomized subjects will have a 4 weeks screening period using NovoRapid® and then 4 weeks treatment period with Fiasp® whereas the rest of the participants will start the trial period with 4 weeks using Fiasp® followed by 4 weeks in NovoRapid®.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained by parents or legal caregivers before any trial-related activities.
2. Any age, age ≥ 2 years and age <18 years at the time of signing informed consent
3. Documented diagnoses of T1DM ≥ 3 months prior to the beginning of the study
4. Using the Medtronic MiniMed 640G system equipped with SmartGuardTM technology and accompanied with EnliteTM Sensor and GuardianTM 2 Link transmitter for at least 30 days prior to beginning of the study and willing to continue using the system throughout the trial.
5. Ability and willingness to use the same insulin infusion sets throughout the trial
6. Using the same insulin for at least 30 days prior to screening
7. HbA1c < 9.0% as assessed by local laboratory at screening
8. Ability and willingness to adhere to the protocol including performing SMBG (Self Monitoring Blood Glucose) profiles, attending visits, uploading pump and sensor data to the CareLink platform

Exclusion Criteria:

1. Participation in another clinical trial within 28 days before the screening visit. Note: clinical trials do not include non-interventional studies
2. Treatment with any medication for the indication of diabetes other than stated in the inclusion criteria within 30 days before screening
3. Anticipated significant change in lifestyle (e.g. eating, exercise or sleeping pattern) throughout the trial
4. Any diabetic complication including renal disease, retinopathy, etc
5. History of hospitalization for ketoacidosis ≤ 3 months prior to the day of screening
6. Any condition which, in the opinion of the Investigator, might influence patient's safety or compliance with the protocol

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-04-15 (Estimated)

PRIMARY OUTCOMES:
1-hour glucose levels on Fiasp | Weeks 1 to 4
  ost-prandial 1-hour glucose levels on Fiasp® when used in the MiniMed 640G pump in children with type 1 diabetes.
1-hour glucose levels on Novorapid | Weeks 1 to 4
  ost-prandial 1-hour glucose levels on Novorapid® when used in the MiniMed 640G pump in children with type 1 diabetes.

SECONDARY OUTCOMES:
Half-hour glucose levels on Fiasp | Weeks 1 to 4
  ost-prandial 1/2-hour glucose levels on Fiasp® when used in the MiniMed
Half-hour glucose levels on Novorapid | Weeks 1 to 4
  ost-prandial 1/2-hour glucose levels on Novorapid® when used in the MiniMed
2 hours glucose levels on Fiasp | Weeks 1 to 4
  ost-prandial 2-hours glucose levels on Fiasp® when used in the MiniMed
2 hours glucose levels on Novorapid | Weeks 1 to 4
  ost-prandial 2-hours glucose levels on Novorapid® when used in the MiniMed
Time in Range in Fiasp | Weeks 1 to 4
  Percent of time spent within 70-180 mg/dl during Fiasp® use
Time in Range in Novorapid | Weeks 1 to 4
  Percent of time spent within 70-180 mg/dl during Novorapid® use
Hypoglycemia in Fiasp | Weeks 1 to 4
  Percent of time spent below 70mg mg/dl during Fiasp® use
Hypoglycemia in Novorapid | Weeks 1 to 4
  Percent of time spent below 70mg mg/dl during Novorapid® use
Total Daily Dose in Fiasp | Weeks 1 to 4
  Units of insulin used per day during Fiasp® use
Total Daily Dose in Novorapid | Weeks 1 to 4
  Units of insulin used per day during Novorapid® use
Basal/Bolus in Fiasp | Weeks 1 to 4
  Units of insulin used per basal/bolus day during Fiasp® use
Basal/Bolus in Novorapid | Weeks 1 to 4
  Units of insulin used per basal/bolus day during Novorapid® use
eHbA1c in Fiasp | Weeks 1 to 4
  Estimated HbA1c levels during Fiasp® use
eHbA1c in Novorapid | Weeks 1 to 4
  Estimated HbA1c levels during Novorapid® use
Incidence of infusion sites reactions in Fiasp | Weeks 1 to 4
  Number of reactions involving infusion sites during Fiasp® use
Incidence of infusion sites reactions in Novorapid | Weeks 1 to 4
  Number of reactions involving infusion sites during Fiasp® use
Occlusion events in Fiasp | Weeks 1 to 4
  Number of occlusion events during Fiasp® use
Occlusion events in Novorapid | Weeks 1 to 4
  Number of occlusion events during Novorapid® use

CONTACTS AND LOCATIONS:
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided